CLINICAL TRIAL: NCT02401425
Title: Use of Letrozole Pretreatment With Misoprostol for First-Trimester Medical Abortion: Randomised Controlled Trial
Brief Title: Use of Letrozole Pretreatment With Misoprostol for First-Trimester Medical Abortion
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Lecturer of obstetrics and gynaecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1984
Record Dates: First submitted 2015-02-25; First posted 2015-03-27 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Complete Miscarriage
Keywords: Letrozole; Misoprostol; First-Trimester; Pretreatment
MeSH Terms: interventions — Letrozole; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- letrozole (Active Comparator): Women will receive three tablets of letrozole(FemaraR, NOVARTIS) as a single dose, each tablet 2.5 mg (total dose 7.5 mg per day) for two days at home and will be told to bring back the empty packs. The third dose will be given on admission to hospital on day three and will be followed by 4 tablets of vaginal misoprostol (200 mcg) (MisotacR,SIGMA)soaked with saline every three hours up to maximum 2 doses.
  Interventions: Drug: Letrozole; Drug: Misoprostol
- placebo (Placebo Comparator): Women will receive three tablets of placebo as a single dose, for two days at home and will be told to bring back the empty packs. The third dose will be given on admission to hospital on day three and will be followed by 4 tablets of vaginal misoprostol (200 mcg) (MisotacR,SIGMA)soaked with saline every three hours up to maximum 2 doses.
  Interventions: Drug: Misoprostol; Other: Placebo

INTERVENTIONS:
Drug: Letrozole
  Other Names: femara
  Arms: letrozole
Drug: Misoprostol
  Other Names: Misotac; Misotec; Cytotec
Other: Placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to compare the success rate of letrozole and misoprostol versus misoprostol alone for medical termination of first trimester pregnancy.

DETAILED DESCRIPTION:
Primary outcome:

Incidence of complete miscarriage (complete expulsion of the products of conception with no need for surgical intervention within one week from the first dose of misoprostol)

Secondary outcome:

Need for surgical evacuation of the products of conception

* Incomplete expulsion of the products of conception (incomplete miscarriage).
* Considerable bleeding necessitating immediate surgical evacuation. Maternal morbidity
* Major side effects (Sepsis, considerable vaginal bleeding leading to hemodynamic instability or necessitating blood transfusion)
* Minor side effects (fever, rigors, nausea, vomiting) Patient's compliance and adherence to treatment Hemoglobin and hematocrit deficit

ELIGIBILITY:
Inclusion Criteria:

* Maternal age more than 18 years old (age of legal consent).
* Gestational age less than 13 weeks.
* Hemoglobin >10 g/dL.
* BMI between 25 kg/m2 and 35 kg/m2.
* Missed abortion.
* Living fetus with multiple congenital malformations incompatible with life.

Exclusion Criteria:

* Maternal age less than 18 years old.
* Gestational age more than 12 weeks.
* Hemoglobin <10 g/dL.
* Anencephaly.
* Fibroid uterus.
* BMI less than 25kg/m2 and more than 35kg/m2.
* Coagulopathy.
* History or evidence of adrenal pathology.
* Previous attempts for induction of abortion in the current pregnancy.
* Allergy to misoprostol or letrozole.
* Medical disorder that contraindicate induction of abortion (e.g. heart failure).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Incidence of complete abortion | 1 week
  complete expulsion of the products of conception with no need for surgical intervention within one week from the first dose of misoprostol

SECONDARY OUTCOMES:
Need for surgical evacuation of the products of conception | 1 week
  Need for surgical evacuation of the products of conception
  * Incomplete expulsion of the products of conception (incomplete miscarriage).
  * Considerable bleeding necessitating immediate surgical evacuation.
Maternal morbidity | 1 week
  Maternal morbidity
  * Major side effects (Sepsis, considerable vaginal bleeding leading to hemodynamic instability or necessitating blood transfusion)
  * Minor side effects (fever, rigors, nausea, vomiting)
Hemoglobin and hematocrit deficit | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt